CLINICAL TRIAL: NCT04047199
Title: Predictive Value of HAS-BLED and CHA2DS2-Vasc Scores for Clinical Outcome After PCI
Brief Title: Predictive Value of HAS-BLED and CHA2DS2-Vasc Scores After PCI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Osama Sayed Morsy, Principal Investigator, Assiut University
Other Study IDs: HAS-BLED-CHA2DS2-Vasc post-PCI
Record Dates: First submitted 2019-08-03; First posted 2019-08-06 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Percutaneous Coronary Intervention
Keywords: Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess the predictive value of two scoring systems, namely HAS-BLED and CHA2DS2-VASc scores, to be linked with bleeding events and recurrence of chest pain and other measures of clinical outcome of percutaneous coronary intervention. The investigators aim to provide evidence for local guidelines of optimum options suited to our population

DETAILED DESCRIPTION:
Dual-antiplatelet therapy (DAPT) with aspirin and an inhibitor of the platelet P2Y12 receptor is necessary to prevent stent-related thrombotic complications after percutaneous coronary intervention (PCI). (1) Although continuation of DAPT confers substantial and durable benefits that extend beyond the local stented segment, bleeding risk also increases with continued exposure to antiplatelet therapy. (2) Current guidelines give fixed duration of DAPT after coronary intervention but many patients still having early stent thrombosis despite this fixed policy, while others, on the contrary, suffer minor and major bleeding events. These clinical situations should raise the possibility of individualizing therapy. (5) The rationale of this study is to find a new method to tailor the optimal duration of DAPT for each patient by balancing long-term risks for both coronary thrombosis and major bleeding (MB).

The HAS-BLED (hypertension, abnormal renal/liver function, stroke, bleeding history or predisposition, labile international normalized ratio, elderly, drugs/alcohol concomitantly) score has long been used to predict bleeding events in patients on anticoagulation therapy. (3) Also, the CHA2DS2-VASc (congestive heart failure, hypertension, ≥75 years, diabetes, stroke/transient ischemic attack or thromboembolism, vascular disease, elderly, sex) score is a well-established system for prediction of thrombo-embolic events in patients with atrial fibrillation. (4) The aim of the present study is to evaluate the predictive ability of these 2 scoring tools when applied to patients undergoing PCI.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing PCI

Exclusion Criteria:

* Those who had undergone unexpected immediate CABG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients who are scheduled for elective PCI (Percutaneous Coronary Intervention) and also those who undergo urgent primary PCI
Sampling Method: Non-Probability Sample
Enrollment: 173 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of bleeding events | 6 months after PCI
  number of bleeding events (epistaxis, bleeding gums, haematuria, GI bleeding, brain bleeding)
Rate of ischaemic events | 6 months after PCI
  number of ischaemic events (ACS, TIA, stroke, acute limb ischaemia, GI, ischaemia)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koene RJ, Win S, Naksuk N, Adatya SN, Rosenbaum AN, John R, Eckman PM. HAS-BLED and CHA(2)DS(2)-VASc scores as predictors of bleeding and thrombotic risk after continuous-flow ventricular assist device implantation. J Card Fail. 2014 Nov;20(11):800-7. doi: 10.1016/j.cardfail.2014.08.010. Epub 2014 Aug 23. PMID 25152496